CLINICAL TRIAL: NCT01791023
Title: The Effect of Acute Exercise on Reactivity and Recovery of Cortisol and DHEAS Levels in Depressive and Healthy Older Adults.
Brief Title: Stress Reactivity of Physical Stressor on Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Helena Sales de Moraes, Principal investigator, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: cortisolexercise01
Record Dates: First submitted 2013-01-04; First posted 2013-02-13 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Depression
Keywords: Depression; Physical exercise; Stress
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical exercise (Experimental): Physical exercise
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — 30 minutes of aerobic exercise on treadmill with moderate intensity.

SUMMARY:
Depressive elderly individuals have showed higher basal level of cortisol and lower level of dehydroepiandrosterone (DHEA). Moreover, changes on these hormone levels have also observed in reactivity of an acute stress, such as physical exercise. On the other hand, physical training can modulate the release of these hormones. Therefore, depressive elderly individuals physically actives might show attenuated reactivity of an acute physical stressor compared to sedentary elderly individuals. The aim of these study is to compare the effect of an acute physical stressor on cortisol levels in depressive and healthy individuals, physically actives and sedentaries. Additionally, the sulfated form of DHEA (DHEAS) serves as a reservoir for DHEA, because of that it is expected that DHEAS levels might reduce after the acute physical exercise.

DETAILED DESCRIPTION:
Depressive and healthy individuals were submitted to one session of 30 minutes of physical exercise of moderate intensity. Before and soon after the exercise it was collected saliva - to analyse cortisol and DHEAS hormones - and some psychological and physical aspects were also collected, such as anamneses, scales of anxiety, temperaments, mood, stress and quality of life. Moreover, during exercise heart rate and mood scale were assessed. To evaluate the reactivity and recovery of physical stressor (physical exercise) saliva tubes and psychological scales were collected 30 minutes and 45 minutes after the end of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age above of 60 years old
* Clinical diagnostic of depression

Exclusion Criteria:

* Hormonal replacement
* Physical disease
* Fasting

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in cortisol and DHEAS levels to after an acute session of exercise | From before and to after one session of 30 minutes of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Helena S Moraes, Ms, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Deolindo Couto Neurology Institute, Rio de Janeiro, Rio de Janeiro, Brazil